CLINICAL TRIAL: NCT05393271
Title: A Randomized, Double-Blind (Sponsor Unblinded), Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Orally Administered VH4011499 in Healthy Participants
Brief Title: First-Time-in-Human (FTIH) Study to Evaluate the Safety, Tolerability and Pharmacokinetics (PK) of VH4011499 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 218490
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections
Keywords: GSK4011499; VH4011499; First-time-in-human; HIV-1 capsid inhibitor; Single ascending doses; Multiple ascending doses; Drug-drug Interaction
MeSH Terms: conditions — HIV Infections | interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: This is a randomized and placebo-controlled study.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind (sponsor unblinded) study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part 1 Single Ascending Dose (SAD): Placebo Powder-in-a-bottle (PiB) (Placebo Comparator): Healthy participants were given a single dose of placebo on Day 1 and were followed up until Day 28.
  Interventions: Drug: Placebo
- Part 1 (SAD): VH4011499 25 mg PiB (Placebo Comparator): Healthy participants were given a single dose of 25 mg VH4011499 on Day 1 and were followed up until Day 28.
  Interventions: Drug: VH4011499
- Part 1 (SAD): VH4011499 125 mg PiB (Experimental): Healthy participants were given a single dose of 125 mg VH4011499 on Day 1 and were followed up until Day 28.
  Interventions: Drug: VH4011499
- Part 1 (SAD): VH4011499 200 mg PiB (Experimental): Healthy participants were given a single dose of 200 mg VH4011499 on Day 1 and were followed up until Day 28.
  Interventions: Drug: VH4011499
- Part 1 (SAD): VH4011499 625 mg PiB (Experimental): Healthy participants were given a single dose of 625 mg VH4011499 on Day 1 and were followed up until Day 28.
  Interventions: Drug: VH4011499
- Part 1 (SAD): VH4011499 1875 mg PiB (Experimental): Healthy participants were given a single dose of 1875 mg VH4011499 on Day 1 and were followed up until Day 28.
  Interventions: Drug: VH4011499
- Part 2 Multiple Ascending Dose (MAD): Placebo PiB (Placebo Comparator): Healthy participants were given a dose of placebo once daily for a 14-day period and were followed up until Day 42.
  Interventions: Drug: Placebo
- Part 2 (MAD): VH4011499 200 mg PiB (Experimental): Healthy participants were given a dose of VH4011499 200 mg PiB once daily for a 14-day period and were followed up until Day 42.
  Interventions: Drug: VH4011499
- Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB (Experimental): Healthy participants were given a dose of VH4011499 300 mg once daily and a single dose of Midazolam on Days 1, 2, and 15, and were followed up until Day 42.
  Interventions: Drug: VH4011499; Drug: Midazolam
- Part 2 (MAD): VH4011499 400 mg PiB (Experimental): Healthy participants were given a dose of VH4011499 400 mg PiB once daily for a 14-day period and were followed up until Day 42.
  Interventions: Drug: VH4011499
- Part 3 (Single dose): VH4011499 200 mg tablet (Experimental): Healthy participants were given a dose of VH4011499 200 mg tablet on Day 1 and were followed up until Day 28.
  Interventions: Drug: VH4011499

INTERVENTIONS:
Drug: VH4011499 — VH4011499 will be administered.
  Other Names: GSK4011499
  Arms: Part 1 (SAD): VH4011499 125 mg PiB; Part 1 (SAD): VH4011499 1875 mg PiB; Part 1 (SAD): VH4011499 200 mg PiB; Part 1 (SAD): VH4011499 25 mg PiB; Part 1 (SAD): VH4011499 625 mg PiB; Part 2 (MAD): VH4011499 200 mg PiB; Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB; Part 2 (MAD): VH4011499 400 mg PiB; Part 3 (Single dose): VH4011499 200 mg tablet
Drug: Placebo — Placebo will be administered.
  Arms: Part 1 Single Ascending Dose (SAD): Placebo Powder-in-a-bottle (PiB); Part 2 Multiple Ascending Dose (MAD): Placebo PiB
Drug: Midazolam — Midazolam will be administered
  Arms: Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB

SUMMARY:
This FTIH study aims to evaluate the safety, tolerability and PK of the novel investigational Human immunodeficiency virus (HIV)-1 capsid inhibitor VH4011499 in healthy adults. The study will be conducted in 3 parts: Part 1 will investigate single ascending doses (SAD) and Part 2 will investigate multiple ascending doses (MAD). Part 3 will investigate single dose of a new formulation of VH4011499. The transition from SAD to MAD will be based on the assessment of the Safety and Dose Escalation Committee.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy.
* Participants must have two consecutive Severe Acute Respiratory Syndrome Coronavirus 2 (SARs-CoV-2) Polymerase chain reaction (PCR) negative results prior to dosing.
* Participants must have body weight > 50 kilograms (kg) and body mass index (BMI) within the range 19-32 kilograms per meter square (kg/m^2).
* Male or female participants (either of non-childbearing potential or of child-bearing potential and using acceptable contraception).
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, neurological or psychiatric disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study drug or interfering with the interpretation of data.
* Abnormal blood pressure.
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) greater than (>)450 milliseconds (msec).
* Past or intended use of over-the-counter or prescription medication including herbal medications within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to dosing and for the duration of the study, unless in the opinion of the Investigator and Sponsor, the medication will not interfere with the study medications, procedures, or compromise participant safety.
* Live vaccine(s) within 1 month prior to screening or plans to receive such vaccines during the study.
* Exposure to more than 4 investigational products within 12 months prior to dosing.
* Current enrollment or recent past participation in another investigational study.
* ALT >1.5 times upper limit of normal (ULN), total bilirubin >1.5 times ULN, and/or estimated serum creatinine clearance less than 60 milliliters per minute.
* History of or current infection with hepatitis B or hepatitis C.
* Positive Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) test, having signs and symptoms, or having contact with known Coronavirus Disease-2019 (COVID-19) positive person/s within 14 days.
* Positive HIV antibody test.
* Use of tobacco or nicotine-containing products, regular alcohol consumption and/or regular use of known drugs of abuse.
* Sensitivity to the study drug, or components thereof midazolam, excipients contained therein, benzodiazepines, or drug or other allergy that, contraindicates participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (2):
- United States (2):
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Study sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf

REFERENCES:
- [Derived] Thakkar N, Griesel R, Pierce A, Bainbridge V, Shepherd B, Angelis K, Tomlinson A, Gandhi Y, Brimhall D, Spears B, Anderson D, Pinnick E, Acuipil C, McCoig C, Baker M, Benn P. Clinical Pharmacokinetics and Safety of Orally Administered VH4011499, a New HIV-1 Capsid Inhibitor, in Adults Without HIV. Infect Dis Ther. 2025 May;14(5):1011-1025. doi: 10.1007/s40121-025-01129-y. Epub 2025 Apr 2. PMID 40172795

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-a-bottle (PiB) | Part 1 (SAD): VH4011499 25 mg PiB | Part 1 (SAD): VH4011499 125 mg PiB | Part 1 (SAD): VH4011499 200 mg PiB | Part 1 (SAD): VH4011499 625 mg PiB | Part 1 (SAD): VH4011499 1875 mg PiB | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4011499 200 mg PiB | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4011499 400 mg PiB | Part 3 (Single Dose): VH4011499 200 mg Tablet
Started | 10 | 6 | 6 | 6 | 6 | 6 | 7 | 6 | 8 | 6 | 6
Completed | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics presented based on Exposed population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-a-bottle (PiB) | Part 1 (SAD): VH4011499 25 mg PiB | Part 1 (SAD): VH4011499 125 mg PiB | Part 1 (SAD): VH4011499 200 mg PiB | Part 1 (SAD): VH4011499 625 mg PiB | Part 1 (SAD): VH4011499 1875 mg PiB | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4011499 200 mg PiB | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4011499 400 mg PiB | Part 3 (Single Dose): VH4011499 200 mg Tablet | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 7 | 6 | 8 | 6 | 6 | 73
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.8 (11.17) | 35.3 (6.12) | 36.5 (7.48) | 45.8 (8.08) | 40.0 (12.05) | 39.8 (7.78) | 37.6 (11.18) | 35.5 (13.10) | 38.9 (11.81) | 32.3 (3.83) | 37.2 (9.91) | 37.9 (9.72)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 9 | 6 | 6 | 5 | 5 | 6 | 7 | 5 | 7 | 6 | 6 | 68
  Female | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 7
  Black or African American | 3 | 3 | 3 | 1 | 2 | 1 | 3 | 3 | 5 | 4 | 1 | 29
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 5 | 2 | 2 | 2 | 4 | 1 | 3 | 3 | 3 | 2 | 3 | 30
  Multiple | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a study intervention whether or not considered related to the study intervention.
Time Frame: Up to Day 28
Population: The analysis was performed on the Safety Set which included all enrolled participants in Part 1 (SAD) who received at least 1 full or partial dose of study treatment. The participants were analyzed according to the treatment they received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-a-bottle (PiB) | Part 1 (SAD): VH4011499 25 mg PiB | Part 1 (SAD): VH4011499 125 mg PiB | Part 1 (SAD): VH4011499 200 mg PiB | Part 1 (SAD): VH4011499 625 mg PiB | Part 1 (SAD): VH4011499 1875 mg PiB
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants | 3 | 2 | 1 | 3 | 1 | 1

2. Primary Outcome: Part 2: Number of Participants With AEs
Description: as for outcome 1
Time Frame: Up to Day 42
Population: The analysis was performed on the Safety Set which included all enrolled participants in Part 2 (MAD) who received at least 1 full or partial dose of study treatment. The participants were analyzed according to the treatment they received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4011499 200 mg PiB | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4011499 400 mg PiB
Number analyzed (Participants) | 7 | 6 | 8 | 6
Participants | 2 | 3 | 3 | 2

3. Primary Outcome: Part 3: Number of Participants With AEs
Description: as for outcome 1
Time Frame: Up to Day 28
Population: The analysis was performed on the Safety Set which included all enrolled participants in Part 3 (Single Dose) who received 1 single dose of study treatment. The participants were analyzed according to the treatment they received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 (Single Dose): VH4011499 200 mg Tablet
Number analyzed (Participants) | 6
Participants | 1

4. Primary Outcome: Part 1: Number of Participants With AEs by Severity
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a study intervention whether or not considered related to the study intervention. The Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric AE was used for all AE severity grading, where Grade 1=Mild symptoms causing no or minimal interference with usual social & functional activities with intervention not indicated, 2=Moderate symptoms causing greater than minimal interference with usual social & functional activities with intervention indicated, 3=Severe symptoms causing inability to perform usual social & functional activities with intervention or hospitalization indicated, 4=Potentially life-threatening symptoms causing inability to perform basic self-care functions with intervention indicated to prevent permanent impairment, persistent disability or death, 5=Death.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-a-bottle (PiB) | Part 1 (SAD): VH4011499 25 mg PiB | Part 1 (SAD): VH4011499 125 mg PiB | Part 1 (SAD): VH4011499 200 mg PiB | Part 1 (SAD): VH4011499 625 mg PiB | Part 1 (SAD): VH4011499 1875 mg PiB
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants
  Grade 1 | 1 | 1 | 1 | 2 | 1 | 1
  Grade 2 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 1 | 0 | 0 | 1 | 0 | 0
  Grade 4 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Part 2: Number of Participants With AEs by Severity
Description: as for outcome 4
Time Frame: Up to Day 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4011499 200 mg PiB | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4011499 400 mg PiB
Number analyzed (Participants) | 7 | 6 | 8 | 6
Participants
  Grade 1 | 2 | 3 | 3 | 2
  Grade 2 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0

6. Primary Outcome: Part 3: Number of Participants With AEs by Severity
Description: as for outcome 4
Time Frame: Up to Day 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 (Single Dose): VH4011499 200 mg Tablet
Number analyzed (Participants) | 6
Participants
  Grade 1 | 1
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

7. Primary Outcome: Part 2: Number of Participants Discontinuing Treatment Due to AEs
Description: Number of participants who discontinued treatment due to AEs are presented.
Time Frame: Up to Day 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4011499 200 mg PiB | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4011499 400 mg PiB
Number analyzed (Participants) | 7 | 6 | 8 | 6
Participants | 0 | 0 | 0 | 0

8. Primary Outcome: Part 1: Absolute Values of Liver Panel Parameters: Direct Bilirubin, Total Bilirubin
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of bilirubin.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micromoles per Liter (μmol/L)
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-a-bottle (PiB) | Part 1 (SAD): VH4011499 25 mg PiB | Part 1 (SAD): VH4011499 125 mg PiB | Part 1 (SAD): VH4011499 200 mg PiB | Part 1 (SAD): VH4011499 625 mg PiB | Part 1 (SAD): VH4011499 1875 mg PiB
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Micromoles per Liter (μmol/L)
  Direct Bilirubin, Baseline (Day 1) | 2.0520 (0.72100) | 2.8500 (1.39621) | 2.2800 (0.88304) | 1.9950 (0.69810) | 2.5650 (0.93661) | 3.1350 (1.28724)
  Direct Bilirubin, Day 2 | 1.9152 (0.88964) | 2.7075 (0.52335) | 1.9950 (0.59891) | 1.9665 (0.49265) | 2.4510 (0.57905) | 3.2205 (1.41183)
  Direct Bilirubin, Day 3 | 1.9665 (0.99465) | 2.5650 (0.64890) | 1.8525 (0.45134) | 1.7385 (0.56628) | 2.3940 (0.66668) | 3.1350 (1.34501)
  Direct Bilirubin, Day 4 | 1.6416 (0.86895) | 2.7075 (0.78300) | 1.9095 (0.48867) | 1.6245 (0.81472) | 2.1375 (0.65562) | 2.7075 (1.01693)
  Direct Bilirubin, Day 5 | 2.0007 (0.75641) | 2.7930 (0.84237) | 2.3085 (0.51584) | 1.7670 (0.35322) | 2.3940 (0.70919) | 3.2205 (1.33519)
  Direct Bilirubin, Day 6 | 1.8639 (0.76239) | 2.8785 (0.95770) | 2.5365 (0.69601) | 1.9380 (0.51490) | 2.2515 (0.63447) | 3.0210 (1.28724)
  Direct Bilirubin, Day 7: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  Direct Bilirubin, Day 7 | 2.1375 (0.84256) | 2.9640 (0.76982) | 2.8044 (0.39367) | 1.6815 (0.67899) | 2.5650 (0.74144) | 3.3630 (1.19292)
  Direct Bilirubin, Day 14: number analyzed (Participants) | 9 | 5 | 6 | 5 | 5 | 6
  Direct Bilirubin, Day 14 | 1.8620 (0.99872) | 2.3256 (1.03027) | 1.9095 (0.64362) | 1.4022 (0.44262) | 1.9494 (0.25933) | 2.0805 (0.93296)
  Direct Bilirubin, Day 21: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Direct Bilirubin, Day 21 | 1.7955 (0.95123) | 2.3256 (0.75123) | 2.1660 (0.50341) | 1.4820 (0.27924) | 1.7385 (0.27396) | 2.2230 (1.08150)
  Direct Bilirubin, Day 28 | 1.7613 (0.75641) | 2.1945 (0.46412) | 1.8810 (0.43260) | 1.7670 (0.45457) | 1.8525 (0.77549) | 2.6220 (1.56226)
  Total Bilirubin, Baseline (Day 1) | 9.4050 (3.14793) | 12.8250 (5.59356) | 10.5450 (4.76555) | 11.6850 (2.27286) | 11.9700 (2.64912) | 13.6800 (6.11788)
  Total Bilirubin, Day 2 | 10.7901 (3.16075) | 11.9415 (2.89069) | 14.0790 (5.31220) | 10.8015 (2.30290) | 13.5945 (3.91997) | 18.5250 (9.28747)
  Total Bilirubin, Day 3 | 10.4310 (2.89748) | 11.9985 (3.02320) | 15.1620 (7.84192) | 11.3145 (2.78980) | 12.5115 (3.76109) | 17.1000 (7.15263)
  Total Bilirubin, Day 4 | 9.6444 (3.82385) | 11.2290 (2.62398) | 12.6825 (6.84634) | 10.1460 (4.36860) | 10.9155 (3.62974) | 15.6465 (7.08175)
  Total Bilirubin, Day 5 | 11.0637 (3.50450) | 12.4260 (2.91938) | 14.6490 (4.95448) | 9.9180 (2.30692) | 12.4545 (3.75331) | 17.7270 (7.77602)
  Total Bilirubin, Day 6 | 10.1574 (3.09505) | 12.3690 (2.20495) | 14.5350 (4.44205) | 10.9725 (2.79189) | 12.1980 (4.57011) | 16.0455 (6.69431)
  Total Bilirubin, Day 7: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  Total Bilirubin, Day 7 | 11.3373 (3.34901) | 13.1670 (3.67391) | 16.1766 (4.75214) | 9.5475 (4.17523) | 12.4545 (4.05153) | 18.1260 (6.43469)
  Total Bilirubin, Day 14: number analyzed (Participants) | 9 | 5 | 6 | 5 | 5 | 6
  Total Bilirubin, Day 14 | 9.1390 (4.16071) | 9.4050 (4.37138) | 9.9750 (3.82011) | 7.5582 (2.48215) | 8.2422 (1.28762) | 10.2885 (4.38563)
  Total Bilirubin, Day 21: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Total Bilirubin, Day 21 | 9.3195 (4.07958) | 9.7128 (2.89793) | 11.0580 (2.83606) | 8.2365 (2.10661) | 8.0370 (1.67894) | 10.5735 (4.85401)
  Total Bilirubin, Day 28 | 9.5247 (3.74733) | 10.4595 (2.49312) | 9.0345 (1.56132) | 9.7185 (2.67858) | 9.1770 (2.78613) | 13.4805 (9.10929)

9. Primary Outcome: Part 1: Absolute Values of Liver Panel Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP) and Aspartate Aminotransferase (AST)
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of ALT, ALP and AST.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: International Units per Liter (IU/L)
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-a-bottle (PiB) | Part 1 (SAD): VH4011499 25 mg PiB | Part 1 (SAD): VH4011499 125 mg PiB | Part 1 (SAD): VH4011499 200 mg PiB | Part 1 (SAD): VH4011499 625 mg PiB | Part 1 (SAD): VH4011499 1875 mg PiB
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
International Units per Liter (IU/L)
  ALP, Baseline (Day 1) | 56.4 (20.82) | 57.2 (18.96) | 53.7 (6.50) | 63.0 (5.14) | 72.0 (29.39) | 55.0 (8.07)
  ALP, Day 2 | 52.3 (17.23) | 56.3 (20.54) | 51.2 (5.34) | 59.3 (5.99) | 67.8 (22.63) | 48.8 (7.05)
  ALP, Day 3 | 53.1 (16.11) | 54.8 (19.36) | 50.7 (6.86) | 58.2 (6.91) | 66.3 (21.08) | 51.7 (8.12)
  ALP, Day 4 | 54.5 (15.63) | 55.5 (19.27) | 52.5 (6.53) | 65.0 (9.82) | 69.5 (24.60) | 52.7 (8.21)
  ALP, Day 5 | 53.9 (14.89) | 54.0 (17.55) | 52.2 (7.22) | 62.2 (9.41) | 68.0 (21.56) | 53.0 (9.34)
  ALP, Day 6 | 54.2 (15.85) | 53.3 (17.45) | 52.3 (8.36) | 65.0 (9.90) | 67.5 (18.72) | 52.7 (9.14)
  ALP, Day 7: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  ALP, Day 7 | 54.6 (15.88) | 54.2 (17.52) | 49.4 (4.56) | 65.0 (10.64) | 66.7 (22.71) | 54.0 (10.00)
  ALP, Day 14: number analyzed (Participants) | 9 | 5 | 6 | 5 | 5 | 6
  ALP, Day 14 | 52.8 (16.59) | 59.6 (24.99) | 53.2 (7.14) | 63.6 (9.71) | 77.2 (22.62) | 53.2 (7.83)
  ALP, Day 21: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  ALP, Day 21 | 58.5 (22.15) | 58.8 (21.48) | 52.8 (6.24) | 66.8 (11.72) | 70.2 (20.49) | 51.3 (6.71)
  ALP, Day 28 | 56.1 (17.62) | 59.0 (19.38) | 55.7 (7.61) | 68.5 (12.14) | 68.7 (20.75) | 51.5 (7.77)
  ALT, Baseline (Day 1) | 13.9 (4.38) | 28.5 (16.01) | 24.7 (9.03) | 16.0 (4.34) | 23.8 (13.11) | 21.7 (3.44)
  ALT, Day 2 | 14.2 (4.96) | 34.0 (24.66) | 23.2 (8.98) | 16.0 (4.98) | 19.5 (10.56) | 21.8 (8.93)
  ALT, Day 3 | 15.7 (5.56) | 33.7 (25.95) | 22.3 (8.04) | 16.5 (5.92) | 17.5 (8.80) | 20.5 (8.48)
  ALT, Day 4 | 16.0 (6.36) | 30.0 (19.93) | 23.2 (7.31) | 15.8 (5.78) | 18.0 (8.72) | 20.3 (7.28)
  ALT, Day 5 | 16.1 (5.36) | 27.2 (16.82) | 22.2 (6.79) | 16.2 (6.11) | 18.2 (9.33) | 19.2 (4.96)
  ALT, Day 6 | 17.4 (6.45) | 24.7 (14.35) | 22.0 (5.44) | 17.2 (6.49) | 17.8 (8.33) | 19.2 (4.49)
  ALT, Day 7: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  ALT, Day 7 | 18.7 (7.56) | 23.5 (12.63) | 23.6 (5.46) | 17.3 (6.53) | 18.2 (9.15) | 20.0 (5.59)
  ALT, Day 14: number analyzed (Participants) | 9 | 5 | 6 | 5 | 5 | 6
  ALT, Day 14 | 19.7 (6.40) | 21.2 (9.50) | 21.5 (6.09) | 16.4 (3.44) | 21.6 (9.24) | 19.7 (3.72)
  ALT, Day 21: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  ALT, Day 21 | 20.5 (11.40) | 26.0 (20.25) | 24.8 (10.55) | 18.2 (3.92) | 19.5 (9.71) | 18.7 (3.61)
  ALT, Day 28 | 24.9 (17.39) | 28.2 (24.81) | 23.8 (6.62) | 16.8 (5.42) | 18.5 (7.48) | 18.2 (3.54)
  AST, Baseline (Day 1) | 15.0 (3.53) | 20.7 (9.65) | 20.3 (3.27) | 16.2 (2.64) | 20.0 (8.07) | 21.7 (4.27)
  AST, Day 2 | 14.2 (3.43) | 23.0 (13.55) | 19.2 (3.66) | 14.3 (3.01) | 15.0 (3.29) | 18.3 (5.57)
  AST, Day 3 | 15.3 (3.16) | 21.0 (9.86) | 18.2 (3.49) | 14.0 (2.37) | 14.7 (2.16) | 17.8 (4.45)
  AST, Day 4 | 15.1 (3.31) | 17.5 (6.83) | 19.3 (3.61) | 14.0 (2.28) | 14.8 (2.64) | 17.8 (3.54)
  AST, Day 5 | 15.2 (2.53) | 15.5 (4.51) | 18.5 (3.02) | 14.2 (2.04) | 14.8 (2.40) | 17.0 (2.76)
  AST, Day 6 | 15.1 (3.41) | 14.8 (3.97) | 18.3 (3.56) | 14.3 (2.07) | 15.0 (1.79) | 17.2 (3.31)
  AST, Day 7: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  AST, Day 7 | 16.0 (3.62) | 17.0 (5.14) | 19.0 (2.55) | 14.7 (2.42) | 14.8 (2.48) | 19.2 (5.19)
  AST, Day 14: number analyzed (Participants) | 9 | 5 | 6 | 5 | 5 | 6
  AST, Day 14 | 18.0 (5.61) | 17.4 (6.66) | 20.7 (5.65) | 17.4 (2.30) | 17.6 (3.21) | 19.5 (4.76)
  AST, Day 21: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  AST, Day 21 | 18.6 (10.07) | 18.4 (6.15) | 20.8 (2.56) | 17.5 (2.07) | 15.8 (3.06) | 19.0 (3.46)
  AST, Day 28 | 20.3 (10.19) | 32.0 (26.50) | 22.8 (5.85) | 15.7 (2.42) | 15.8 (2.71) | 19.8 (4.49)

10. Primary Outcome: Part 2: Absolute Values of Liver Panel Parameters: Direct Bilirubin, Total Bilirubin
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of bilirubin.
Time Frame: Up to Day 42
Population: The analysis was performed on the Safety Set which included all enrolled participants in Part 2 (MAD) who received at least 1 full or partial dose of study treatment. The participants were analyzed according to the treatment they received. Only those participants with data available at the specified timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4011499 200 mg PiB | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4011499 400 mg PiB
Number analyzed (Participants) | 7 | 6 | 8 | 6
μmol/L
  Direct Bilirubin, Baseline (Day 1) | 1.6856 (0.34805) | 1.7670 (0.88304) | 1.6031 (0.74782) | 2.5365 (1.12089)
  Direct Bilirubin, Day 2: number analyzed (Participants) | 5 | 6 | 0 | 6
  Direct Bilirubin, Day 2 | 1.8126 (0.35459) | 1.9665 (0.66448) |  | 2.8785 (1.15177)
  Direct Bilirubin, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 3 | 1.8810 (0.24183) |  | 2.1161 (0.56298) |
  Direct Bilirubin, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 5 | 1.9238 (0.64551) | 2.3370 (0.71466) |  | 2.4510 (0.75447)
  Direct Bilirubin, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 6 | 1.8810 (0.24183) |  | 2.4795 (0.60630) |
  Direct Bilirubin, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 7 | 2.1375 (0.40706) | 2.0805 (0.81949) |  | 3.2490 (1.23310)
  Direct Bilirubin, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 8 | 1.6245 (0.36275) |  | 2.2444 (0.43296) |
  Direct Bilirubin, Day 11: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 11 | 2.1803 (0.56499) | 2.1660 (0.62752) |  | 3.1065 (1.18678)
  Direct Bilirubin, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 12 | 1.3680 (0.24183) |  | 2.2871 (0.48312) |
  Direct Bilirubin, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 14 | 2.1375 (0.45242) | 2.1660 (0.61813) |  | 3.0495 (1.15683)
  Direct Bilirubin, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 15 | 1.9665 (0.12092) |  | 2.2444 (0.37058) |
  Direct Bilirubin, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 21 | 1.9665 (0.35596) | 1.9950 (0.61813) |  | 2.8785 (1.17190)
  Direct Bilirubin, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 22 | 1.7955 (0.36275) |  | 2.0734 (0.58838) |
  Direct Bilirubin, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  Direct Bilirubin, Day 28 | 1.5048 (0.38994) | 1.3965 (0.58657) | 1.2825 (0.44778) | 1.8525 (0.76026)
  Direct Bilirubin, Day 35: number analyzed (Participants) | 6 | 6 | 8 | 6
  Direct Bilirubin, Day 35 | 1.4250 (0.33625) | 1.4535 (0.49265) | 1.3253 (0.27037) | 2.8500 (1.72927)
  Direct Bilirubin, Day 42: number analyzed (Participants) | 6 | 6 | 8 | 6
  Direct Bilirubin, Day 42 | 1.5105 (0.36542) | 1.1115 (0.50438) | 1.7100 (0.34200) | 2.5650 (1.97947)
  Total Bilirubin, Baseline (Day 1) | 10.5776 (2.98545) | 10.0890 (5.90780) | 9.5760 (4.36923) | 12.8250 (6.63163)
  Total Bilirubin, Day 2: number analyzed (Participants) | 5 | 6 | 0 | 6
  Total Bilirubin, Day 2 | 12.1752 (1.75806) | 13.6800 (6.64924) |  | 16.8720 (7.08416)
  Total Bilirubin, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 3 | 12.1410 (1.69281) |  | 12.5044 (4.14193) |
  Total Bilirubin, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 5 | 12.0128 (2.81458) | 13.7370 (5.74282) |  | 15.7320 (4.92171)
  Total Bilirubin, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 6 | 10.0890 (1.93464) |  | 12.7181 (3.00651) |
  Total Bilirubin, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 7 | 12.8250 (2.43837) | 13.2240 (6.58176) |  | 16.4445 (6.72047)
  Total Bilirubin, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 8 | 9.9180 (1.69281) |  | 13.1456 (2.44141) |
  Total Bilirubin, Day 11: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 11 | 12.7395 (2.48392) | 13.8510 (5.61547) |  | 16.4445 (6.63464)
  Total Bilirubin, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 12 | 10.6875 (0.36275) |  | 13.8724 (4.15402) |
  Total Bilirubin, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 14 | 11.7563 (2.12378) | 13.4235 (4.72994) |  | 15.6465 (6.66132)
  Total Bilirubin, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 15 | 11.7990 (2.66014) |  | 13.9793 (3.89270) |
  Total Bilirubin, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 21 | 12.5258 (0.21517) | 11.9700 (4.29070) |  | 16.9575 (7.40445)
  Total Bilirubin, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 22 | 11.2005 (2.29739) |  | 12.2479 (3.78959) |
  Total Bilirubin, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  Total Bilirubin, Day 28 | 8.5842 (2.34276) | 8.1225 (4.03031) | 6.6904 (2.71983) | 8.3220 (3.44499)
  Total Bilirubin, Day 35: number analyzed (Participants) | 6 | 6 | 8 | 6
  Total Bilirubin, Day 35 | 9.1770 (2.04534) | 8.2365 (2.28761) | 7.5454 (2.29136) | 15.0195 (10.22140)
  Total Bilirubin, Day 42: number analyzed (Participants) | 6 | 6 | 8 | 6
  Total Bilirubin, Day 42 | 9.7755 (3.14643) | 7.4385 (2.67712) | 8.6141 (2.36934) | 13.0530 (11.74742)

11. Primary Outcome: Part 2: Absolute Values of Liver Panel Parameters: ALT, ALP and AST
Description: as for outcome 9
Time Frame: Up to Day 42
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4011499 200 mg PiB | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4011499 400 mg PiB
Number analyzed (Participants) | 7 | 6 | 8 | 6
IU/L
  ALP, Baseline (Day 1) | 56.0 (16.78) | 59.5 (19.69) | 69.0 (22.43) | 53.8 (10.55)
  ALP, Day 2: number analyzed (Participants) | 5 | 6 | 0 | 6
  ALP, Day 2 | 53.8 (12.15) | 58.3 (20.97) |  | 53.2 (10.91)
  ALP, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 3 | 47.0 (18.38) |  | 68.6 (22.56) |
  ALP, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 5 | 52.5 (10.34) | 62.2 (23.59) |  | 54.3 (11.04)
  ALP, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 6 | 47.0 (18.38) |  | 69.3 (21.99) |
  ALP, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 7 | 50.3 (12.04) | 59.3 (20.65) |  | 54.2 (10.46)
  ALP, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 8 | 47.0 (18.38) |  | 71.9 (24.31) |
  ALP, Day 11: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 11 | 50.3 (12.92) | 54.0 (18.07) |  | 51.2 (9.77)
  ALP, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 12 | 47.0 (18.38) |  | 64.0 (19.95) |
  ALP, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 14 | 51.8 (12.76) | 61.0 (19.78) |  | 49.7 (9.20)
  ALP, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 15 | 50.5 (23.33) |  | 66.5 (22.60) |
  ALP, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 21 | 49.5 (12.40) | 51.8 (14.30) |  | 50.8 (10.53)
  ALP, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 22 | 47.0 (18.38) |  | 63.8 (18.72) |
  ALP, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  ALP, Day 28 | 53.4 (11.67) | 60.0 (14.85) | 62.6 (19.26) | 51.3 (10.67)
  ALP, Day 35: number analyzed (Participants) | 6 | 6 | 8 | 6
  ALP, Day 35 | 47.7 (12.71) | 63.0 (34.89) | 65.5 (17.88) | 49.0 (11.37)
  ALP, Day 42: number analyzed (Participants) | 6 | 6 | 8 | 6
  ALP, Day 42 | 52.2 (12.64) | 60.3 (18.60) | 66.5 (22.53) | 53.5 (10.65)
  ALT, Baseline (Day 1) | 23.6 (8.30) | 15.8 (4.62) | 19.5 (5.71) | 19.8 (6.24)
  ALT, Day 2: number analyzed (Participants) | 5 | 6 | 0 | 6
  ALT, Day 2 | 19.8 (6.30) | 16.0 (4.90) |  | 19.0 (6.03)
  ALT, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 3 | 23.5 (12.02) |  | 16.6 (4.47) |
  ALT, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 5 | 17.0 (5.35) | 16.0 (4.65) |  | 17.3 (6.31)
  ALT, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 6 | 19.5 (9.19) |  | 15.6 (5.48) |
  ALT, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 7 | 16.0 (4.24) | 14.5 (3.62) |  | 18.8 (7.47)
  ALT, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 8 | 20.5 (7.78) |  | 18.1 (7.86) |
  ALT, Day 11: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 11 | 15.3 (3.77) | 12.5 (3.73) |  | 19.5 (8.76)
  ALT, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 12 | 18.0 (8.49) |  | 14.8 (5.85) |
  ALT, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 14 | 16.8 (4.19) | 12.2 (3.19) |  | 18.7 (7.31)
  ALT, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 15 | 26.0 (16.97) |  | 18.1 (7.75) |
  ALT, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 21 | 16.0 (5.35) | 12.3 (3.33) |  | 18.3 (8.19)
  ALT, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 22 | 19.5 (10.61) |  | 17.0 (8.72) |
  ALT, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  ALT, Day 28 | 20.6 (9.29) | 16.7 (6.02) | 20.9 (7.59) | 22.3 (11.41)
  ALT, Day 35: number analyzed (Participants) | 6 | 6 | 8 | 6
  ALT, Day 35 | 22.0 (11.76) | 28.0 (27.79) | 18.4 (5.93) | 18.3 (4.13)
  ALT, Day 42: number analyzed (Participants) | 6 | 6 | 8 | 6
  ALT, Day 42 | 24.2 (10.38) | 14.8 (3.66) | 20.5 (5.93) | 21.8 (4.45)
  AST, Baseline (Day 1) | 23.3 (7.45) | 17.3 (3.44) | 18.9 (2.70) | 17.7 (3.27)
  AST, Day 2: number analyzed (Participants) | 5 | 6 | 0 | 6
  AST, Day 2 | 19.6 (2.61) | 16.5 (3.02) |  | 15.3 (3.08)
  AST, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 3 | 19.0 (8.49) |  | 17.0 (2.98) |
  AST, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 5 | 18.0 (2.83) | 16.8 (2.04) |  | 14.0 (2.10)
  AST, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 6 | 16.0 (7.07) |  | 16.0 (3.07) |
  AST, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 7 | 17.3 (1.71) | 16.3 (2.25) |  | 14.7 (1.63)
  AST, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 8 | 17.0 (5.66) |  | 18.0 (4.69) |
  AST, Day 11: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 11 | 15.5 (2.38) | 15.8 (3.54) |  | 13.3 (2.50)
  AST, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 12 | 16.5 (4.95) |  | 15.9 (2.70) |
  AST, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 14 | 17.3 (3.10) | 16.7 (3.50) |  | 13.8 (2.14)
  AST, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 15 | 20.0 (9.90) |  | 17.6 (4.17) |
  AST, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 21 | 16.5 (2.08) | 15.7 (2.73) |  | 15.0 (3.16)
  AST, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 22 | 18.0 (4.24) |  | 16.6 (3.16) |
  AST, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  AST, Day 28 | 20.2 (4.27) | 17.5 (3.73) | 22.6 (8.19) | 20.7 (7.84)
  AST, Day 35: number analyzed (Participants) | 6 | 6 | 8 | 6
  AST, Day 35 | 20.0 (6.63) | 26.3 (19.34) | 20.5 (3.55) | 20.2 (7.91)
  AST, Day 42: number analyzed (Participants) | 6 | 6 | 8 | 6
  AST, Day 42 | 21.7 (4.93) | 16.3 (1.75) | 19.8 (4.20) | 20.7 (3.27)

12. Primary Outcome: Part 3: Absolute Values of Liver Panel Parameters: Direct Bilirubin, Total Bilirubin
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of bilirubin.
Time Frame: Up to Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part 3 (Single Dose): VH4011499 200 mg Tablet
Number analyzed (Participants) | 6
IU/L
  Direct Bilirubin, Baseline (Day 1) | 1.4250 (0.69810)
  Direct Bilirubin, Day 2 | 2.1375 (0.97784)
  Direct Bilirubin, Day 3 | 2.2515 (1.05642)
  Direct Bilirubin, Day 4 | 1.9665 (0.94747)
  Direct Bilirubin, Day 5: number analyzed (Participants) | 5
  Direct Bilirubin, Day 5 | 1.7784 (0.44591)
  Direct Bilirubin, Day 6 | 2.3085 (1.11216)
  Direct Bilirubin, Day 7 | 1.9950 (0.89619)
  Direct Bilirubin, Day 14 | 1.9665 (0.69038)
  Direct Bilirubin, Day 21 | 1.8525 (0.69601)
  Direct Bilirubin, Day 28 | 2.6790 (2.39074)
  Total Bilirubin, Baseline (Day 1) | 7.6950 (3.19912)
  Total Bilirubin, Day 2 | 14.2500 (7.57873)
  Total Bilirubin, Day 3 | 13.8225 (7.43283)
  Total Bilirubin, Day 4 | 12.2550 (6.56575)
  Total Bilirubin, Day 5: number analyzed (Participants) | 5
  Total Bilirubin, Day 5 | 10.8756 (2.84755)
  Total Bilirubin, Day 6 | 14.5920 (8.80586)
  Total Bilirubin, Day 7 | 11.2290 (5.55123)
  Total Bilirubin, Day 14 | 11.7705 (6.12879)
  Total Bilirubin, Day 21 | 8.2365 (3.08827)
  Total Bilirubin, Day 28 | 14.4495 (15.05412)

13. Primary Outcome: Part 3: Absolute Values of Liver Panel Parameters: ALT, ALP and AST
Description: as for outcome 9
Time Frame: Up to Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Part 3 (Single Dose): VH4011499 200 mg Tablet
Number analyzed (Participants) | 6
μmol/L
  ALP, Baseline (Day 1) | 52.0 (8.12)
  ALP, Day 2 | 50.7 (7.99)
  ALP, Day 3 | 51.0 (8.20)
  ALP, Day 4 | 54.3 (7.39)
  ALP, Day 5: number analyzed (Participants) | 5
  ALP, Day 5 | 56.6 (7.73)
  ALP, Day 6 | 54.2 (6.62)
  ALP, Day 7 | 54.7 (6.12)
  ALP, Day 14 | 54.7 (10.39)
  ALP, Day 21 | 52.7 (7.61)
  ALP, Day 28 | 56.3 (8.52)
  ALT, Baseline (Day 1) | 12.7 (4.03)
  ALT, Day 2 | 15.2 (6.74)
  ALT, Day 3 | 15.0 (6.60)
  ALT, Day 4 | 15.0 (8.32)
  ALT, Day 5: number analyzed (Participants) | 5
  ALT, Day 5 | 13.0 (4.42)
  ALT, Day 6 | 15.2 (6.85)
  ALT, Day 7 | 15.0 (5.87)
  ALT, Day 14 | 17.5 (8.96)
  ALT, Day 21 | 19.2 (10.26)
  ALT, Day 28 | 15.0 (4.38)
  AST, Baseline | 16.7 (1.63)
  AST, Day 2 | 17.3 (3.20)
  AST, Day 3 | 16.3 (2.34)
  AST, Day 4 | 16.5 (2.26)
  AST, Day 5: number analyzed (Participants) | 5
  AST, Day 5 | 16.6 (1.14)
  AST, Day 6 | 17.2 (1.83)
  AST, Day 7 | 16.3 (1.63)
  AST, Day 14 | 19.3 (3.44)
  AST, Day 21 | 21.0 (9.03)
  AST, Day 28 | 18.5 (3.27)

14. Primary Outcome: Part 1: Change From Baseline in Liver Panel Parameters: Direct Bilirubin, Total Bilirubin
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of bilirubin. Change from baseline was calculated by subtracting the baseline value from the post-dose visit value.
Time Frame: From Baseline (Day 1) and up to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-a-bottle (PiB) | Part 1 (SAD): VH4011499 25 mg PiB | Part 1 (SAD): VH4011499 125 mg PiB | Part 1 (SAD): VH4011499 200 mg PiB | Part 1 (SAD): VH4011499 625 mg PiB | Part 1 (SAD): VH4011499 1875 mg PiB
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
IU/L
  Direct Bilirubin, Baseline (Day 1) | 2.0520 (0.72100) | 2.8500 (1.39621) | 2.2800 (0.88304) | 1.9950 (0.69810) | 2.5650 (0.93661) | 3.1350 (1.28724)
  Direct Bilirubin, Day 2 | -0.1368 (0.54553) | -0.1425 (1.54248) | -0.2850 (0.84237) | -0.0285 (0.45134) | -0.1140 (0.62752) | 0.0855 (0.79289)
  Direct Bilirubin, Day 3 | -0.0855 (0.99465) | -0.2850 (1.53963) | -0.4275 (0.90968) | -0.2565 (0.35459) | -0.1710 (0.78734) | 0.0000 (1.14965)
  Direct Bilirubin, Day 4 | -0.4104 (0.49822) | -0.1425 (1.53868) | -0.3705 (0.90754) | -0.3705 (0.62518) | -0.4275 (0.55936) | -0.4275 (0.84985)
  Direct Bilirubin, Day 5 | -0.0513 (0.58157) | -0.0570 (1.84384) | 0.0285 (1.02267) | -0.2280 (0.73085) | -0.1710 (0.66668) | 0.0855 (1.00148)
  Direct Bilirubin, Day 6 | -0.1881 (0.49331) | 0.0285 (2.01872) | 0.2565 (1.30117) | -0.0570 (0.56886) | -0.3135 (0.63447) | -0.1140 (1.30976)
  Direct Bilirubin, Day 7: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  Direct Bilirubin, Day 7 | 0.0855 (0.56571) | 0.1140 (1.77928) | 0.4104 (1.00148) | -0.3135 (0.47656) | 0.0000 (0.61179) | 0.2280 (1.21719)
  Direct Bilirubin, Day 14: number analyzed (Participants) | 9 | 5 | 6 | 5 | 5 | 6
  Direct Bilirubin, Day 14 | -0.2280 (0.61655) | -0.4104 (1.21277) | -0.3705 (1.11040) | -0.6498 (0.89999) | -0.7866 (0.98678) | -1.0545 (1.05087)
  Direct Bilirubin, Day 21: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Direct Bilirubin, Day 21 | -0.2565 (0.50502) | -0.4104 (1.12523) | -0.1140 (1.09047) | -0.5130 (0.72549) | -0.8265 (0.88138) | -0.9120 (0.97735)
  Direct Bilirubin, Day 28 | -0.2907 (0.39532) | -0.6555 (1.80457) | -0.3990 (0.98331) | -0.2280 (0.70643) | -0.7125 (0.77549) | -0.5130 (1.16982)
  Total Bilirubin, Baseline (Day 1) | 9.4050 (3.14793) | 12.8250 (5.59356) | 10.5450 (4.76555) | 11.6850 (2.27286) | 11.9700 (2.64912) | 13.6800 (6.11788)
  Total Bilirubin, Day 2 | 1.3851 (2.24764) | -0.8835 (4.85401) | 3.5340 (4.59817) | -0.8835 (2.06171) | 1.6245 (2.72261) | 4.8450 (6.74934)
  Total Bilirubin, Day 3 | 1.0260 (2.05042) | -0.8265 (5.51609) | 4.6170 (7.54418) | -0.3705 (1.79482) | 0.5415 (2.92088) | 3.4200 (7.47252)
  Total Bilirubin, Day 4 | 0.2394 (2.41185) | -1.5960 (5.05381) | 2.1375 (6.66747) | -1.5390 (3.11577) | -1.0545 (2.33568) | 1.9665 (5.79158)
  Total Bilirubin, Day 5 | 1.6587 (2.37773) | -0.3990 (5.95676) | 4.1040 (5.26169) | -1.7670 (2.50541) | 0.4845 (1.97774) | 4.0470 (7.46913)
  Total Bilirubin, Day 6 | 0.7524 (2.27886) | -0.4560 (6.19451) | 3.9900 (6.70064) | -0.7125 (1.83031) | 0.2280 (3.36078) | 2.3655 (8.26581)
  Total Bilirubin, Day 7: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  Total Bilirubin, Day 7 | 1.9323 (2.55682) | 0.3420 (6.36984) | 5.2326 (5.27972) | -2.1375 (2.49859) | 0.4845 (2.42655) | 4.4460 (6.95867)
  Total Bilirubin, Day 14: number analyzed (Participants) | 9 | 5 | 6 | 5 | 5 | 6
  Total Bilirubin, Day 14 | -0.3610 (1.91460) | -2.9070 (6.29108) | -0.5700 (4.06486) | -4.0698 (3.91698) | -3.7278 (3.46966) | -3.3915 (4.65725)
  Total Bilirubin, Day 21: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Total Bilirubin, Day 21 | -0.0855 (2.10399) | -2.5992 (5.51776) | 0.5130 (3.87835) | -3.4485 (2.88056) | -3.9330 (2.82228) | -3.1065 (3.89102)
  Total Bilirubin, Day 28 | 0.1197 (1.42169) | -2.3655 (7.17501) | -1.5105 (4.15838) | -1.9665 (3.32770) | -2.7930 (2.63510) | -0.1995 (5.55096)

15. Primary Outcome: Part 1: Change From Baseline in Liver Panel Parameters: ALT, ALP and AST
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of ALT, ALP and AST. Change from baseline was calculated by subtracting the baseline value from the post-dose visit value.
Time Frame: From Baseline (Day 1) and up to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-a-bottle (PiB) | Part 1 (SAD): VH4011499 25 mg PiB | Part 1 (SAD): VH4011499 125 mg PiB | Part 1 (SAD): VH4011499 200 mg PiB | Part 1 (SAD): VH4011499 625 mg PiB | Part 1 (SAD): VH4011499 1875 mg PiB
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
μmol/L
  ALP, Baseline (Day 1) | 56.4 (20.82) | 57.2 (18.96) | 53.7 (6.50) | 63.0 (5.14) | 72.0 (29.39) | 55.0 (8.07)
  ALP, Day 2 | -4.1 (6.35) | -0.8 (3.13) | -2.5 (3.27) | -3.7 (3.50) | -4.2 (7.41) | -6.2 (2.71)
  ALP, Day 3 | -3.3 (6.00) | -2.3 (3.39) | -3.0 (5.06) | -4.8 (4.02) | -5.7 (9.37) | -3.3 (3.39)
  ALP, Day 4 | -1.9 (7.74) | -1.7 (3.39) | -1.2 (5.19) | 2.0 (6.39) | -2.5 (7.48) | -2.3 (2.73)
  ALP, Day 5 | -2.5 (7.35) | -3.2 (4.07) | -1.5 (4.09) | -0.8 (5.98) | -4.0 (9.27) | -2.0 (3.46)
  ALP, Day 6 | -2.2 (7.07) | -3.8 (3.54) | -1.3 (5.43) | 2.0 (6.42) | -4.5 (12.88) | -2.3 (3.39)
  ALP, Day 7: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  ALP, Day 7 | -1.8 (8.01) | -3.0 (4.20) | -3.2 (4.32) | 2.0 (6.63) | -5.3 (9.77) | -1.0 (3.16)
  ALP, Day 14: number analyzed (Participants) | 9 | 5 | 6 | 5 | 5 | 6
  ALP, Day 14 | 0.4 (5.77) | 0.8 (8.58) | -0.5 (5.75) | 0.0 (5.15) | 0.0 (7.35) | -1.8 (3.13)
  ALP, Day 21: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  ALP, Day 21 | 2.1 (12.14) | 0.0 (4.90) | -0.8 (3.19) | 3.8 (8.40) | -1.8 (11.48) | -3.7 (3.44)
  ALP, Day 28 | -0.3 (7.06) | 1.8 (3.87) | 2.0 (8.72) | 5.5 (8.48) | -3.3 (9.40) | -3.5 (3.56)
  ALT, Baseline (Day 1) | 13.9 (4.38) | 28.5 (16.01) | 24.7 (9.03) | 16.0 (4.34) | 23.8 (13.11) | 21.7 (3.44)
  ALT, Day 2 | 0.3 (1.89) | 5.5 (11.26) | -1.5 (3.39) | 0.0 (1.55) | -4.3 (3.78) | 0.2 (7.19)
  ALT, Day 3 | 1.8 (2.44) | 5.2 (13.04) | -2.3 (3.08) | 0.5 (2.43) | -6.3 (5.20) | -1.2 (7.14)
  ALT, Day 4 | 2.1 (3.87) | 1.5 (6.02) | -1.5 (4.28) | -0.2 (2.23) | -5.8 (5.64) | -1.3 (6.47)
  ALT, Day 5 | 2.2 (3.49) | -1.3 (3.72) | -2.5 (3.73) | 0.2 (2.48) | -5.7 (6.35) | -2.5 (5.21)
  ALT, Day 6 | 3.5 (4.97) | -3.8 (3.87) | -2.7 (5.54) | 1.2 (3.19) | -6.0 (7.72) | -2.5 (5.39)
  ALT, Day 7: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  ALT, Day 7 | 4.8 (5.96) | -5.0 (5.37) | -3.6 (5.41) | 1.3 (2.73) | -5.7 (7.45) | -1.7 (6.71)
  ALT, Day 14: number analyzed (Participants) | 9 | 5 | 6 | 5 | 5 | 6
  ALT, Day 14 | 5.3 (5.48) | -7.0 (9.41) | -3.2 (4.45) | 0.8 (2.17) | -1.0 (6.16) | -2.0 (5.18)
  ALT, Day 21: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  ALT, Day 21 | 6.6 (8.78) | -2.2 (13.50) | 0.2 (8.40) | 2.2 (3.60) | -4.3 (6.89) | -3.0 (4.47)
  ALT, Day 28 | 11.0 (17.58) | -0.3 (15.47) | -0.8 (4.12) | 0.8 (3.19) | -5.3 (8.85) | -3.5 (2.43)
  AST, Baseline (Day 1) | 15.0 (3.53) | 20.7 (9.65) | 20.3 (3.27) | 16.2 (2.64) | 20.0 (8.07) | 21.7 (4.27)
  AST, Day 2 | -0.8 (1.32) | 2.3 (9.03) | -1.2 (2.04) | -1.8 (1.83) | -5.0 (5.44) | -3.3 (4.84)
  AST, Day 3 | 0.3 (2.54) | 0.3 (6.35) | -2.2 (1.94) | -2.2 (2.64) | -5.3 (6.83) | -3.8 (4.31)
  AST, Day 4 | 0.1 (2.33) | -3.2 (3.76) | -1.0 (2.10) | -2.2 (2.32) | -5.2 (6.62) | -3.8 (4.02)
  AST, Day 5 | 0.2 (2.44) | -5.2 (5.56) | -1.8 (0.75) | -2.0 (2.28) | -5.2 (6.88) | -4.7 (3.27)
  AST, Day 6 | 0.1 (2.18) | -5.8 (6.11) | -2.0 (2.10) | -1.8 (2.64) | -5.0 (7.24) | -4.5 (3.21)
  AST, Day 7: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  AST, Day 7 | 1.0 (3.16) | -3.7 (7.84) | -2.0 (1.58) | -1.5 (2.17) | -5.2 (7.08) | -2.5 (3.78)
  AST, Day 14: number analyzed (Participants) | 9 | 5 | 6 | 5 | 5 | 6
  AST, Day 14 | 2.7 (5.79) | -3.6 (5.03) | 0.3 (2.88) | 0.8 (0.84) | -3.0 (6.28) | -2.2 (4.96)
  AST, Day 21: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  AST, Day 21 | 3.6 (7.57) | -2.6 (6.11) | 0.5 (4.51) | 1.3 (2.34) | -4.2 (5.78) | -2.7 (2.73)
  AST, Day 28 | 5.3 (8.63) | 11.3 (17.81) | 2.5 (4.28) | -0.5 (2.43) | -4.2 (7.44) | -1.8 (3.19)

16. Primary Outcome: Part 2: Change From Baseline in Liver Panel Parameters: Direct Bilirubin, Total Bilirubin
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of bilirubin. Change from baseline was calculated by subtracting the baseline value from the post-dose visit value. Standard Deviation (SD)=0.0000 is defined as following: if all participants analyzed for a specific parameter at a specific time point have the same value, then SD is equal with 0.0000.
Time Frame: From Baseline (Day 1) and up to Day 42
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4011499 200 mg PiB | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4011499 400 mg PiB
Number analyzed (Participants) | 7 | 6 | 8 | 6
μmol/L
  Direct Bilirubin, Baseline (Day 1) | 1.6856 (0.34805) | 1.7670 (0.88304) | 1.6031 (0.74782) | 2.5365 (1.12089)
  Direct Bilirubin, Day 2: number analyzed (Participants) | 5 | 6 | 0 | 6
  Direct Bilirubin, Day 2 | 0.1368 (0.67756) | 0.1995 (0.43820) |  | 0.3420 (0.32445)
  Direct Bilirubin, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 3 | 0.1710 (0.0000) |  | 0.5130 (0.35400) |
  Direct Bilirubin, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 5 | 0.2565 (1.04948) | 0.5700 (0.42807) |  | -0.0855 (0.44262)
  Direct Bilirubin, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 6 | 0.1710 (0.0000) |  | 0.8764 (0.54412) |
  Direct Bilirubin, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 7 | 0.4703 (0.76950) | 0.3135 (0.36542) |  | 0.7125 (0.36542)
  Direct Bilirubin, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 8 | -0.0855 (0.12092) |  | 0.6413 (0.60458) |
  Direct Bilirubin, Day 11: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 11 | 0.5130 (0.91556) | 0.3990 (0.31838) |  | 0.5700 (0.46726)
  Direct Bilirubin, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 12 | -0.3420 (0.0000) |  | 0.6840 (0.48366) |
  Direct Bilirubin, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 14 | 0.4703 (0.66044) | 0.3990 (0.36940) |  | 0.5130 (0.30589)
  Direct Bilirubin, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 15 | 0.2565 (0.12092) |  | 0.6413 (0.42628) |
  Direct Bilirubin, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  Direct Bilirubin, Day 21 | 0.2993 (0.78206) | 0.2280 (0.46726) |  | 0.3420 (0.35869)
  Direct Bilirubin, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  Direct Bilirubin, Day 22 | 0.0855 (0.12092) |  | 0.4703 (0.53881) |
  Direct Bilirubin, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  Direct Bilirubin, Day 28 | -0.2052 (0.77800) | -0.3705 (0.52335) | -0.3206 (0.57401) | -0.6840 (0.71739)
  Direct Bilirubin, Day 35: number analyzed (Participants) | 6 | 6 | 8 | 6
  Direct Bilirubin, Day 35 | -0.2565 (0.44262) | -0.3135 (0.61576) | -0.2779 (0.56298) | 0.3135 (0.75253)
  Direct Bilirubin, Day 42: number analyzed (Participants) | 6 | 6 | 8 | 6
  Direct Bilirubin, Day 42 | -0.1710 (0.37464) | -0.6555 (0.46412) | 0.1069 (0.63942) | 0.0285 (0.89456)
  Total Bilirubin, Baseline (Day 1) | 10.5776 (2.98545) | 10.0890 (5.90780) | 9.5760 (4.36923) | 12.8250 (6.63163)
  Total Bilirubin, Day 2: number analyzed (Participants) | 5 | 6 | 0 | 6
  Total Bilirubin, Day 2 | 2.0520 (4.88623) | 3.5910 (1.49466) |  | 4.0470 (1.90622)
  Total Bilirubin, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 3 | 0.4275 (0.12092) |  | 2.9284 (1.86301) |
  Total Bilirubin, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 5 | 1.3253 (6.24774) | 3.6480 (1.09582) |  | 2.9070 (2.52478)
  Total Bilirubin, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 6 | -1.6245 (0.36275) |  | 3.1421 (2.90044) |
  Total Bilirubin, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 7 | 2.1375 (5.96052) | 3.1350 (2.20495) |  | 3.6195 (1.75529)
  Total Bilirubin, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 8 | -1.7955 (0.12092) |  | 3.5696 (3.25149) |
  Total Bilirubin, Day 11: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 11 | 2.0520 (5.83575) | 3.7620 (2.69508) |  | 3.6195 (1.29517)
  Total Bilirubin, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 12 | -1.0260 (1.20915) |  | 4.2964 (2.74733) |
  Total Bilirubin, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 14 | 1.0688 (4.14271) | 3.3345 (1.83138) |  | 2.8215 (1.26932)
  Total Bilirubin, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 15 | 0.0855 (1.08824) |  | 4.4033 (2.53263) |
  Total Bilirubin, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  Total Bilirubin, Day 21 | 1.8383 (3.83481) | 1.8810 (3.11577) |  | 4.1325 (2.32816)
  Total Bilirubin, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  Total Bilirubin, Day 22 | -0.5130 (0.72549) |  | 2.6719 (3.49125) |
  Total Bilirubin, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  Total Bilirubin, Day 28 | -2.5308 (5.31257) | -1.9665 (3.28525) | -2.8856 (2.53212) | -4.5030 (4.18257)
  Total Bilirubin, Day 35: number analyzed (Participants) | 6 | 6 | 8 | 6
  Total Bilirubin, Day 35 | -1.8525 (3.35337) | -1.8525 (4.50534) | -2.0306 (2.42251) | 2.1945 (4.64845)
  Total Bilirubin, Day 42: number analyzed (Participants) | 6 | 6 | 8 | 6
  Total Bilirubin, Day 42 | -1.2540 (2.32376) | -2.6505 (4.28354) | -0.9619 (3.56231) | 0.2280 (5.78644)

17. Primary Outcome: Part 2: Change From Baseline in Liver Panel Parameters: ALT, ALP and AST
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of ALT, ALP and AST. Change from baseline was calculated by subtracting the baseline value from the post-dose visit value. SD=0.00 is defined as following: if all participants analyzed for a specific parameter at a specific time point have the same value, then SD is equal with 0.00.
Time Frame: From Baseline (Day 1) and up to Day 42
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4011499 200 mg PiB | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4011499 400 mg PiB
Number analyzed (Participants) | 7 | 6 | 8 | 6
IU/L
  ALP, Baseline (Day 1) | 56.0 (16.78) | 59.5 (19.69) | 69.0 (22.43) | 53.8 (10.55)
  ALP, Day 2: number analyzed (Participants) | 5 | 6 | 0 | 6
  ALP, Day 2 | -5.8 (12.48) | -1.2 (3.92) |  | -0.7 (3.50)
  ALP, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 3 | 0.0 (1.41) |  | -0.4 (2.20) |
  ALP, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 5 | -6.8 (14.31) | 2.7 (5.09) |  | 0.5 (2.59)
  ALP, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 6 | 0.0 (1.41) |  | 0.3 (3.41) |
  ALP, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 7 | -9.0 (14.31) | -0.2 (3.66) |  | 0.3 (3.33)
  ALP, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 8 | 0.0 (1.41) |  | 2.9 (7.32) |
  ALP, Day 11: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 11 | -9.0 (16.02) | -5.5 (3.89) |  | -2.7 (4.08)
  ALP, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 12 | 0.0 (1.41) |  | -5.0 (3.34) |
  ALP, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 14 | -7.5 (15.15) | 1.5 (3.56) |  | -4.2 (3.60)
  ALP, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 15 | 3.5 (3.54) |  | -2.5 (3.70) |
  ALP, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALP, Day 21 | -9.8 (15.59) | -7.7 (6.44) |  | -3.0 (4.82)
  ALP, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALP, Day 22 | 0.0 (1.41) |  | -5.3 (5.63) |
  ALP, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  ALP, Day 28 | -6.2 (11.23) | 0.5 (9.52) | -6.4 (4.96) | -2.5 (3.15)
  ALP, Day 35: number analyzed (Participants) | 6 | 6 | 8 | 6
  ALP, Day 35 | -7.5 (7.79) | 3.5 (17.16) | -3.5 (6.21) | -4.8 (1.83)
  ALP, Day 42: number analyzed (Participants) | 6 | 6 | 8 | 6
  ALP, Day 42 | -3.0 (7.48) | 0.8 (8.08) | -2.5 (3.63) | -0.3 (3.72)
  ALT, Baseline (Day 1) | 23.6 (8.30) | 15.8 (4.62) | 19.5 (5.71) | 19.8 (6.24)
  ALT, Day 2: number analyzed (Participants) | 5 | 6 | 0 | 6
  ALT, Day 2 | -2.6 (2.41) | 0.2 (1.72) |  | -0.8 (2.32)
  ALT, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 3 | -3.0 (1.41) |  | -2.9 (3.56) |
  ALT, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 5 | -4.5 (4.20) | 0.2 (2.64) |  | -2.5 (2.74)
  ALT, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 6 | -7.0 (1.41) |  | -3.9 (5.82) |
  ALT, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 7 | -5.5 (5.74) | -1.3 (2.07) |  | -1.0 (2.97)
  ALT, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 8 | -6.0 (2.83) |  | -1.4 (8.58) |
  ALT, Day 11: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 11 | -6.3 (6.02) | -3.3 (3.67) |  | -0.3 (5.47)
  ALT, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 12 | -8.5 (2.12) |  | -4.8 (7.19) |
  ALT, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 14 | -4.8 (5.85) | -3.7 (4.46) |  | -1.2 (3.66)
  ALT, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 15 | -0.5 (6.36) |  | -1.4 (8.85) |
  ALT, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  ALT, Day 21 | -5.5 (4.65) | -3.5 (4.04) |  | -1.5 (5.47)
  ALT, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  ALT, Day 22 | -7.0 (0.00) |  | -2.5 (9.43) |
  ALT, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  ALT, Day 28 | -3.4 (7.09) | 0.8 (3.66) | 1.4 (5.78) | 2.5 (8.46)
  ALT, Day 35: number analyzed (Participants) | 6 | 6 | 8 | 6
  ALT, Day 35 | -1.2 (8.47) | 12.2 (25.97) | -1.1 (4.26) | -1.5 (4.51)
  ALT, Day 42: number analyzed (Participants) | 6 | 6 | 8 | 6
  ALT, Day 42 | 1.0 (8.39) | -1.0 (4.29) | 1.0 (2.45) | 2.0 (4.10)
  AST, Baseline (Day 1) | 23.3 (7.45) | 17.3 (3.44) | 18.9 (2.70) | 17.7 (3.27)
  AST, Day 2: number analyzed (Participants) | 5 | 6 | 0 | 6
  AST, Day 2 | -4.4 (5.81) | -0.8 (1.47) |  | -2.3 (2.25)
  AST, Day 3: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 3 | -2.5 (0.71) |  | -1.9 (2.23) |
  AST, Day 5: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 5 | -2.5 (1.00) | -0.5 (1.87) |  | -3.7 (2.73)
  AST, Day 6: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 6 | -5.5 (0.71) |  | -2.9 (3.14) |
  AST, Day 7: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 7 | -3.3 (1.89) | -1.0 (2.10) |  | -3.0 (2.45)
  AST, Day 8: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 8 | -4.5 (2.12) |  | -0.9 (4.29) |
  AST, Day 11: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 11 | -5.0 (3.16) | -1.5 (1.64) |  | -4.3 (3.01)
  AST, Day 12: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 12 | -5.0 (2.83) |  | -3.0 (2.45) |
  AST, Day 14: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 14 | -3.3 (2.22) | -0.7 (2.73) |  | -3.8 (2.32)
  AST, Day 15: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 15 | -1.5 (2.12) |  | -1.3 (3.81) |
  AST, Day 21: number analyzed (Participants) | 4 | 6 | 0 | 6
  AST, Day 21 | -4.0 (1.83) | -1.7 (2.25) |  | -2.7 (3.83)
  AST, Day 22: number analyzed (Participants) | 2 | 0 | 8 | 0
  AST, Day 22 | -3.5 (3.54) |  | -2.3 (3.20) |
  AST, Day 28: number analyzed (Participants) | 5 | 6 | 8 | 6
  AST, Day 28 | -1.6 (3.13) | 0.2 (2.56) | 3.8 (9.08) | 3.0 (5.73)
  AST, Day 35: number analyzed (Participants) | 6 | 6 | 8 | 6
  AST, Day 35 | -0.8 (4.54) | 9.0 (19.07) | 1.6 (3.81) | 2.5 (5.96)
  AST, Day 42: number analyzed (Participants) | 6 | 6 | 8 | 6
  AST, Day 42 | 0.8 (5.34) | -1.0 (2.61) | 0.9 (3.44) | 3.0 (5.33)

18. Primary Outcome: Part 3: Change From Baseline in Liver Panel Parameters: Direct Bilirubin, Total Bilirubin
Description: as for outcome 14
Time Frame: From Baseline (Day 1) and up to Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part 3 (Single Dose): VH4011499 200 mg Tablet
Number analyzed (Participants) | 6
IU/L
  Direct Bilirubin, Baseline (Day 1) | 1.4250 (0.69810)
  Direct Bilirubin, Day 2 | 0.7125 (0.89456)
  Direct Bilirubin, Day 3 | 0.8265 (0.93920)
  Direct Bilirubin, Day 4 | 0.5415 (0.92667)
  Direct Bilirubin, Day 5: number analyzed (Participants) | 5
  Direct Bilirubin, Day 5 | 0.4104 (0.53531)
  Direct Bilirubin, Day 6 | 0.8835 (0.98182)
  Direct Bilirubin, Day 7 | 0.5700 (0.79228)
  Direct Bilirubin, Day 14 | 0.5415 (0.66154)
  Direct Bilirubin, Day 21 | 0.4275 (0.41536)
  Direct Bilirubin, Day 28 | 1.2540 (2.25219)
  Total Bilirubin, Baseline (Day 1) | 7.6950 (3.19912)
  Total Bilirubin, Day 2 | 6.5550 (6.58354)
  Total Bilirubin, Day 3 | 6.1275 (6.16873)
  Total Bilirubin, Day 4 | 4.5600 (5.75401)
  Total Bilirubin, Day 5: number analyzed (Participants) | 5
  Total Bilirubin, Day 5 | 3.6936 (3.29058)
  Total Bilirubin, Day 6 | 6.8970 (7.58181)
  Total Bilirubin, Day 7 | 3.5340 (5.11821)
  Total Bilirubin, Day 14 | 4.0755 (4.44786)
  Total Bilirubin, Day 21 | 0.5415 (2.47901)
  Total Bilirubin, Day 28 | 6.7545 (13.42355)

19. Primary Outcome: Part 3: Change From Baseline in Liver Panel Parameters: ALT, ALP and AST
Description: as for outcome 15
Time Frame: From Baseline (Day 1) and up to Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part 3 (Single Dose): VH4011499 200 mg Tablet
Number analyzed (Participants) | 6
IU/L
  ALP, Baseline (Day 1) | 52.0 (8.12)
  ALP, Day 2 | -1.3 (6.02)
  ALP, Day 3 | -1.0 (6.29)
  ALP, Day 4 | 2.3 (6.31)
  ALP, Day 5: number analyzed (Participants) | 5
  ALP, Day 5 | 5.4 (5.73)
  ALP, Day 6 | 2.2 (6.52)
  ALP, Day 7 | 2.7 (6.47)
  ALP, Day 14 | 2.7 (7.17)
  ALP, Day 21 | 0.7 (6.02)
  ALP, Day 28 | 4.3 (5.50)
  ALT, Baseline (Day 1) | 12.7 (4.03)
  ALT, Day 2 | 2.5 (5.17)
  ALT, Day 3 | 2.3 (5.57)
  ALT, Day 4 | 2.3 (6.98)
  ALT, Day 5: number analyzed (Participants) | 5
  ALT, Day 5 | 0.8 (1.64)
  ALT, Day 6 | 2.5 (4.42)
  ALT, Day 7 | 2.3 (3.39)
  ALT, Day 14 | 4.8 (5.60)
  ALT, Day 21 | 6.5 (6.66)
  ALT, Day 28 | 2.3 (1.03)
  AST, Baseline (Day 1) | 16.7 (1.63)
  AST, Day 2 | 0.7 (3.50)
  AST, Day 3 | -0.3 (2.34)
  AST, Day 4 | -0.2 (2.64)
  AST, Day 5: number analyzed (Participants) | 5
  AST, Day 5 | -0.4 (1.52)
  AST, Day 6 | 0.5 (1.87)
  AST, Day 7 | -0.3 (1.86)
  AST, Day 14 | 2.7 (3.27)
  AST, Day 21 | 4.3 (7.79)
  AST, Day 28 | 1.8 (2.56)

20. Primary Outcome: Part 1: Number of Participants With Maximum Toxicity Grade Increase From Baseline for Liver Panel Parameters
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of the liver panel parameters: ALT, ALP, AST, total bilirubin and direct bilirubin. The number of participants with any grade increase (from grade 1 [mild] to grade 4 [potentially life-threatening]) have been presented.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-a-bottle (PiB) | Part 1 (SAD): VH4011499 25 mg PiB | Part 1 (SAD): VH4011499 125 mg PiB | Part 1 (SAD): VH4011499 200 mg PiB | Part 1 (SAD): VH4011499 625 mg PiB | Part 1 (SAD): VH4011499 1875 mg PiB
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants
  ALT, Increase to Grade 1 | 0 | 2 | 0 | 0 | 0 | 0
  ALT, Increase to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Increase to Grade 1 | 0 | 2 | 0 | 0 | 0 | 0
  AST, Increase to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

21. Primary Outcome: Part 2: Number of Participants With Maximum Toxicity Grade Increase From Baseline for Liver Panel Parameters
Description: as for outcome 20
Time Frame: Up to Day 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4011499 200 mg PiB | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4011499 400 mg PiB
Number analyzed (Participants) | 7 | 6 | 8 | 6
Participants
  ALT, Increase to Grade 1 | 0 | 1 | 0 | 0
  ALT, Increase to Grade 2 | 0 | 0 | 0 | 0
  ALT, Increase to Grade 3 | 0 | 0 | 0 | 0
  ALT, Increase to Grade 4 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 1 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 2 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 3 | 0 | 0 | 0 | 0
  ALP, Increase to Grade 4 | 0 | 0 | 0 | 0
  AST, Increase to Grade 1 | 0 | 1 | 0 | 0
  AST, Increase to Grade 2 | 0 | 0 | 0 | 0
  AST, Increase to Grade 3 | 0 | 0 | 0 | 0
  AST, Increase to Grade 4 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 1 | 0 | 0 | 0 | 1
  Total Bilirubin, Increase to Grade 2 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 3 | 0 | 0 | 0 | 0
  Total Bilirubin, Increase to Grade 4 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 1 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 2 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 3 | 0 | 0 | 0 | 0
  Direct Bilirubin, Increase to Grade 4 | 0 | 0 | 0 | 0

22. Primary Outcome: Part 3: Number of Participants With Maximum Toxicity Grade Increase From Baseline for Liver Panel Parameters
Description: as for outcome 20
Time Frame: Up to Day 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 (Single Dose): VH4011499 200 mg Tablet
Number analyzed (Participants) | 6
Participants
  ALT, Increase to Grade 1 | 0
  ALT, Increase to Grade 2 | 0
  ALT, Increase to Grade 3 | 0
  ALT, Increase to Grade 4 | 0
  ALP, Increase to Grade 1 | 0
  ALP, Increase to Grade 2 | 0
  ALP, Increase to Grade 3 | 0
  ALP, Increase to Grade 4 | 0
  AST, Increase to Grade 1 | 0
  AST, Increase to Grade 2 | 0
  AST, Increase to Grade 3 | 0
  AST, Increase to Grade 4 | 0
  Total Bilirubin, Increase to Grade 1 | 1
  Total Bilirubin, Increase to Grade 2 | 0
  Total Bilirubin, Increase to Grade 3 | 0
  Total Bilirubin, Increase to Grade 4 | 0
  Direct Bilirubin, Increase to Grade 1 | 0
  Direct Bilirubin, Increase to Grade 2 | 0
  Direct Bilirubin, Increase to Grade 3 | 0
  Direct Bilirubin, Increase to Grade 4 | 0

23. Primary Outcome: Part 1: Area Under the Plasma Concentration Time Curve (AUC) From Time Zero to Infinity (0-inf) Following Single Dose Administration of VH4011499
Description: Blood samples were collected as assessed by protocol, at specific time points for pharmacokinetic (PK) analysis to determine AUC(0-inf). For AUC, a linear trapezoidal method was employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method was used for those arising from decreasing concentrations. Geometric Coefficient of Variation was expressed in percentages.
Time Frame: At Day 1
Population: The analysis was performed on the VH4011499 PK Set which included all participants in the Part 1 (SAD) Safety Set who received at least 1 full dose of study treatment with at least one non-missing PK assessment. The participants were analyzed according to the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour nanogram per milliliter (h*ng/mL)
Arm/Group | Part 1 (SAD): VH4011499 25 mg PiB | Part 1 (SAD): VH4011499 125 mg PiB | Part 1 (SAD): VH4011499 200 mg PiB | Part 1 (SAD): VH4011499 625 mg PiB | Part 1 (SAD): VH4011499 1875 mg PiB
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Hour nanogram per milliliter (h*ng/mL) | 2759.51 (53.69) | 8458.88 (20.39) | 11627.63 (36.01) | 24391.58 (34.16) | 36327.28 (48.29)

24. Primary Outcome: Part 2: AUC Over a Dosing Interval From Time of Dosing to the Time of the Subsequent Dose (0-t) Following Repeat Dose Administration of VH4011499
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis to determine AUC(0-t). For AUC, a linear trapezoidal method was employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method was used for those arising from decreasing concentrations.
Time Frame: At Days 1 and 14 for Part 2 (MAD): VH4011499 200 mg PiB and Part 2 (MAD): VH4011499 400 mg PiB groups, and at Days 2 and 15 for Part 2 (MAD): VH4011499 300 mg + Midazolam PiB group
Population: The analysis was performed on the VH4011499 PK Set which included all participants in the Part 2 (MAD) Safety Set who received at least 1 full dose of study treatment with at least one non-missing PK assessment. The participants were analyzed according to the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 2 (MAD): VH4011499 200 mg PiB | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4011499 400 mg PiB
Number analyzed (Participants) | 6 | 8 | 6
h*ng/mL
  Day 1/2 | 4211.67 (15.36) | 5385.19 (21.74) | 4879.14 (36.00)
  Day 14/15 | 95735.06 (56.77) | 168459.8 (54.17) | 139259.6 (24.66)

25. Primary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) Following Single Dose Administration of VH4011499.
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis to determine Cmax.
Time Frame: At Day 1
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1 (SAD): VH4011499 25 mg PiB | Part 1 (SAD): VH4011499 125 mg PiB | Part 1 (SAD): VH4011499 200 mg PiB | Part 1 (SAD): VH4011499 625 mg PiB | Part 1 (SAD): VH4011499 1875 mg PiB
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL) | 26.85 (26.18) | 106.90 (17.24) | 168.88 (36.25) | 328.95 (37.97) | 557.81 (52.86)

26. Primary Outcome: Part 1: Time to Maximum Observed Plasma Concentration (Tmax) Following Single Dose Administration of VH4011499
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis to determine Tmax.
Time Frame: At Day 1
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1 (SAD): VH4011499 25 mg PiB | Part 1 (SAD): VH4011499 125 mg PiB | Part 1 (SAD): VH4011499 200 mg PiB | Part 1 (SAD): VH4011499 625 mg PiB | Part 1 (SAD): VH4011499 1875 mg PiB
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hours | 11.30 (9.51) | 10.26 (14.77) | 9.28 (11.56) | 7.86 (22.83) | 8.79 (24.60)

27. Primary Outcome: Part 1: Apparent Terminal Half-life (T1/2) Following Single Dose Administration of VH4011499
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis to determine T1/2.
Time Frame: At Day 1
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1 (SAD): VH4011499 25 mg PiB | Part 1 (SAD): VH4011499 125 mg PiB | Part 1 (SAD): VH4011499 200 mg PiB | Part 1 (SAD): VH4011499 625 mg PiB | Part 1 (SAD): VH4011499 1875 mg PiB
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hours | 63.97 (21.07) | 54.44 (23.86) | 61.61 (29.57) | 66.32 (24.75) | 55.90 (25.33)

28. Primary Outcome: Part 2: Cmax Following Repeat Dose Administration of VH4011499
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis to determine Cmax.
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2 (MAD): VH4011499 200 mg PiB | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4011499 400 mg PiB
Number analyzed (Participants) | 6 | 8 | 6
ng/mL
  Day 1: number analyzed (Participants) | 6 | 0 | 6
  Day 1 | 260.89 (19.62) |  | 321.37 (53.14)
  Day 2: number analyzed (Participants) | 0 | 8 | 0
  Day 2 |  | 348.24 (20.46) |
  Day 14: number analyzed (Participants) | 6 | 0 | 6
  Day 14 | 1272.25 (42.47) |  | 1509.90 (22.56)
  Day 15: number analyzed (Participants) | 0 | 8 | 0
  Day 15 |  | 1913.76 (22.93) |

29. Primary Outcome: Part 2: Tmax Following Repeat Dose Administration of VH4011499
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis to determine Tmax.
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2 (MAD): VH4011499 200 mg PiB | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4011499 400 mg PiB
Number analyzed (Participants) | 6 | 8 | 6
hours
  Day 1: number analyzed (Participants) | 6 | 0 | 6
  Day 1 | 10.71 (41.53) |  | 9.50 (51.00)
  Day 2: number analyzed (Participants) | 0 | 8 | 0
  Day 2 |  | 8.11 (22.96) |
  Day 14: number analyzed (Participants) | 6 | 0 | 6
  Day 14 | 4.80 (30.46) |  | 5.99 (42.79)
  Day 15: number analyzed (Participants) | 0 | 8 | 0
  Day 15 |  | 5.27 (32.11) |

30. Primary Outcome: Part 2: T1/2 Following Repeat Dose Administration of VH4011499
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis to determine T1/2.
Time Frame: At Day 14 for Part 2 (MAD): VH4011499 200 mg PiB and Part 2 (MAD): VH4011499 400 mg PiB groups, and at Day 15 for Part 2 (MAD): VH4011499 300 mg + Midazolam PiB group
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2 (MAD): VH4011499 200 mg PiB | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4011499 400 mg PiB
Number analyzed (Participants) | 6 | 8 | 6
hours
  Day 14: number analyzed (Participants) | 6 | 0 | 6
  Day 14 | 51.17 (16.68) |  | 60.36 (21.81)
  Day 15: number analyzed (Participants) | 0 | 8 | 0
  Day 15 |  | 66.47 (19.10) |

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events and serious adverse events were collected up to 28-days following final dose of VH4011499 or placebo (Day 28 for Part 1 and Part 3, and Day 42 for Part 2).
Description: The analysis was performed on the Safety Set which included all participants who received at least 1 full or partial dose of study treatment.
Arm/Group | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-a-bottle (PiB) | Part 1 (SAD): VH4011499 25 mg PiB | Part 1 (SAD): VH4011499 125 mg PiB | Part 1 (SAD): VH4011499 200 mg PiB | Part 1 (SAD): VH4011499 625 mg PiB | Part 1 (SAD): VH4011499 1875 mg PiB | Part 2 Multiple Ascending Dose (MAD): Placebo PiB | Part 2 (MAD): VH4011499 200 mg PiB | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB | Part 2 (MAD): VH4011499 400 mg PiB | Part 3 (Single Dose): VH4011499 200 mg Tablet
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/8 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/8 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/10 | 2/6 | 1/6 | 3/6 | 1/6 | 1/6 | 2/7 | 3/6 | 3/8 | 2/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-a-bottle (PiB) (N=10) | Part 1 (SAD): VH4011499 25 mg PiB (N=6) | Part 1 (SAD): VH4011499 125 mg PiB (N=6) | Part 1 (SAD): VH4011499 200 mg PiB (N=6) | Part 1 (SAD): VH4011499 625 mg PiB (N=6) | Part 1 (SAD): VH4011499 1875 mg PiB (N=6) | Part 2 Multiple Ascending Dose (MAD): Placebo PiB (N=7) | Part 2 (MAD): VH4011499 200 mg PiB (N=6) | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB (N=8) | Part 2 (MAD): VH4011499 400 mg PiB (N=6) | Part 3 (Single Dose): VH4011499 200 mg Tablet (N=6)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Single Ascending Dose (SAD): Placebo Powder-in-a-bottle (PiB) (N=10) | Part 1 (SAD): VH4011499 25 mg PiB (N=6) | Part 1 (SAD): VH4011499 125 mg PiB (N=6) | Part 1 (SAD): VH4011499 200 mg PiB (N=6) | Part 1 (SAD): VH4011499 625 mg PiB (N=6) | Part 1 (SAD): VH4011499 1875 mg PiB (N=6) | Part 2 Multiple Ascending Dose (MAD): Placebo PiB (N=7) | Part 2 (MAD): VH4011499 200 mg PiB (N=6) | Part 2 (MAD): VH4011499 300 mg + Midazolam (MDZ) PiB (N=8) | Part 2 (MAD): VH4011499 400 mg PiB (N=6) | Part 3 (Single Dose): VH4011499 200 mg Tablet (N=6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site dermatitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Total bile acids increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT05393271/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT05393271/SAP_001.pdf